CLINICAL TRIAL: NCT06535984
Title: The Effect of White Noise and Swaddling on Pain, Heart Rate, and Oxygen Saturation in Term İnfants Undergoing Eye Examinations: A Randomised Controlled Trial
Brief Title: The Effect of White Noise and Swaddling on Pain, Heart Rate, and Oxygen Saturation in Term İnfants Undergoing Eye Examinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Sultan GÜNER BAŞARA, Erbaa Faculty of Health Sciences, Department of Nursing, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Tokat Gaziosmanpaşa University
Record Dates: First submitted 2024-07-05; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Pain
Keywords: Eye examination; İnfant; Pain; Nonpharmacologic
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants were divided into four groups: three intervention groups and one control group. Infants were assigned to these groups using simple random sampling to ensure homogeneity and prevent selection bias. The sample size was calculated using the G-Power 3.0.10 program. With a confidence interval (CI) of 95%, α = 0.05, effect size = 0.159, and power (1 - β) = 0.80, a total sample size of 108 was calculated for the four groups, with at least 27 infants in each group. The study included 120 infants divided into the swaddling group (n=30), white noise group (n=30), white noise + swaddling group (n=30), and control group (n=30)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In the data collection process, the person collecting data was not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- white noise (Experimental): In the research, white noise was provided to the experimental group
  Interventions: Other: White Noise
- swaddling (Experimental): In the research, swaddling was provided to the experimental group
  Interventions: Other: Swaddling
- White Noise + Swaddling group (Experimental): In the research, White Noise + Swaddling group were provided to the experimental group
  Interventions: Other: White Noise+Swaddling
- Control group (No Intervention): The control group received routine care

INTERVENTIONS:
Other: White Noise — White Noise Group (n=30) The third researcher turned on white noise (rain sound; link: https://www.youtube.com/watch?v=rZeM-HZeneo) before the start of the eye examination and played it to the infants until the end of the examination.
  Arms: white noise
Other: Swaddling — Swaddling group (n=30) The third researcher swaddled each infant with its thin blanket. The swaddling involved bringing the infant's left hand close to the left buttock and wrapping it with the upper right end of the blanket. Similarly, she wrapped the baby's right hand with the upper left end of the blanket by bringing it closer to the right hip. She wrapped the baby's legs with the lower part of the blanket, ensuring that the baby's head could move freely.
  Arms: swaddling
Other: White Noise+Swaddling — White Noise + Swaddling Group (n=30) The third researcher swaddled the infants in this group as described in the swaddling group and turned on the white noise (rain sound; link: https://www.youtube.com/watch?v=rZeM-HZeneo) before the examination started and played it to the infants until the examination was over.
  Arms: White Noise + Swaddling group

SUMMARY:
Eye examinations for vision screening in infants cause pain and stress. Aim: To evaluate the effect of white noise and swaddling on pain, heart rate, and oxygen saturation in term infants undergoing post-discharge eye examinations. This study was conducted with term infants born 30-36 days postpartum who visited the ophthalmologic outpatient clinic for eye screening. A total of 120 term infants were included in the sample, divided into three intervention groups: the white noise group (n=30), the swaddling group (n=30), and the white noise + swaddling group (n=30), along with a control group (n=30). Data were collected by the clinic nurse before the eye examination, 30 seconds into the examination, and at the end of the examination. The Premature Infant Pain Profile (PIPP) scale and pulse oximetry were used for data collection.There was no statistically significant difference in pain scores, heart rates, or oxygen saturation (SpO2) between the intervention and control groups (p>0.05). In all groups, pain scores and heart rates were higher, and SpO2 values were lower after the ophthalmologic examination than before the examination (p<0.001).Swaddling + white noise, white noise, and swaddling during the eye examination procedure did not affect reducing infants' pain or improving heart rate and oxygen saturation values.

DETAILED DESCRIPTION:
Early childhood is a critical period for identifying and treating eye diseases, as problems that develop during this time can lead to permanent vision loss. It is recommended that term infants be evaluated for congenital cataracts, congenital glaucoma, retinoblastoma, strabismus, amblyopia, and refractive errors. An estimated 20,000-40,000 babies are born with bilateral cataracts each year globally, leading to blindness in over 14 million children. Congenital glaucoma, a developmental disorder that can be unilateral or bilateral, often occurs at birth or within the first few months of life and can damage the optic nerve, leading to vision loss. The incidence of congenital glaucoma in developed countries is approximately 1 in 10,000-20,000 births. Infections such as rubella and cytomegalovirus (CMV) during pregnancy can also cause cataracts and glaucoma in infants. Detecting risk factors that could impede normal vision development through infant vision screening and providing early treatment helps prevent vision loss and blindness. In Turkey, the national vision screening program includes routine eye examinations and red reflex tests conducted by family physicians for infants aged 0-3 years. Additionally, term infants who do not require intensive care undergo detailed examinations for eye diseases like congenital cataracts and glaucoma at two reference hospitals designated by the Ministry of Health. These examinations use similar methods to those employed in retinopathy of prematurity (RP) screening.

Eye examinations for screening and early diagnosis can be painful and stressful for infants. Exposure to pain can lead to hypersensitivity to painful stimuli, a decreased pain threshold, and altered cortex development in the short term, as well as long-term behavioral problems and learning difficulties. Therefore, it is crucial to minimize pain and stress during these examinations. Systemic pharmacological analgesics used to reduce pain in infants can negatively impact their early brain development, nutrition, socialization, and memory in later years. Currently, non-pharmacologic methods to reduce pain in infants are gaining prominence. These methods are more cost-effective, easier to administer, and safer compared to pharmacologic approaches. They can also be used in combination with pharmacologic treatments. Various non-pharmacological methods frequently used for analgesia in newborns and infants include kangaroo care, swaddling, non-nutritive sucking, exposure to specific odors (such as from the mother, breast milk, or aromatic scents), sucrose, glucose, breast milk, music therapy, massage, white noise, and acupuncture. During eye examinations, blefastop is used to keep the baby's eyelids open, and a scleral depressor is employed to assess the bottom of the eye and move the eye sideways, causing discomfort. The white light source used by the ophthalmologist further unsettles the baby. Studies have explored different non-pharmacologic methods to reduce pain during eye examinations in premature infants, including touch, positioning, non-nutritive sucking, breast milk, glucose, sucrose, white noise, and music. However, these studies have yielded conflicting results, and the evidence remains insufficient. Upon reviewing the literature, no studies were encountered comparing the effects of non-pharmacologic methods on reducing pain during eye examinations in term infants. There is a need for further research to investigate the effectiveness of non-pharmacologic methods in alleviating pain during post-discharge eye examinations in term infants.

This study aimed to evaluate the effect of white noise and swaddling on interventional pain, heart rate, and oxygen saturation (SpO2) in term infants undergoing hospital eye examinations for post-discharge vision screening.

Hypotheses of the Study:

H01: Playing white noise to babies during eye examinations does not affect pain scores, heart rate, or oxygen saturation.

H02: Swaddling infants during eye examinations does not affect pain scores, heart rate, or oxygen saturation.

H03: Swaddling combined with listening to white noise during eye examinations does not affect pain scores, heart rate, or oxygen saturation.

Methods This study was a prospective, randomized, controlled experimental study. The study was conducted in the neonatal eye outpatient clinic of a maternity hospital.In this hospital, healthy infants who do not require intensive care after birth are given screening eye examinations once between the 30th and 36th days after birth. Approximately 400 infants who do not need intensive care are admitted to the neonatal eye outpatient clinic each month. Participants were divided into four groups: three intervention groups and one control group. Infants were assigned to these groups using simple random sampling to ensure homogeneity and prevent selection bias. The sample size was calculated using the G-Power 3.0.10 program. With a confidence interval (CI) of 95%, α = 0.05, effect size = 0.159, and power (1 - β) = 0.80, a total sample size of 108 was calculated for the four groups, with at least 27 infants in each group. The study included 120 infants divided into the swaddling group (n=30), white noise group (n=30), white noise + swaddling group (n=30), and control group (n=30) (Figure 1). The sample included infants with a gestational age of >37 6/7 weeks, birth weight ≥2000 g, a 5th minute Apgar score ≥7, aged 30-36 days postpartum, and undergoing their first eye examination. The exclusion criteria included a history of hospitalization in the neonatal intensive care unit, postnatal resuscitation, presence or suspicion of a congenital and/or genetic disease, hearing problems, surgical operation for any reason, or systemic analgesic administration within the last six hours. No infants dropped out of the study during the study period.Interventions Infants who were swaddled during the eye examination constituted the swaddling group (Intervention Group-1). Infants who listened to white noise constituted the white noise group (Intervention Group-2). Infants who were both swaddled and listened to white noise during the eye examination constituted the White Noise + Swaddling group (Intervention Group-3). The control group received routine care and follow-up. The outpatient clinic nurse (third researcher) numbered the babies according to their order of admission and assigned them to groups by simple randomization. All infants were examined by the same ophthalmologist (fourth investigator). Another outpatient nurse, who was not part of the research team, measured the infants' pain scores, heart rate, and oxygen saturation at three different times: before the examination (T1), 30 seconds after the ophthalmologist started the first eye examination (T2), and immediately after the examination of the second eye was finished (T3).

Eye Examination Preparation: All infants included in the study (intervention groups 1, 2, and 3, as well as the control group) underwent routine procedures performed in the eye outpatient clinic before the examination. During this stage, pupil dilation was initiated in the waiting room. According to the hospital's standard procedure, the pupil dilation process involved instilling phenylephrine and tropicamide eye drops twice at five-minute intervals (Liu et al., 2017). Approximately 45 minutes later, once the pupils were dilated, each infant was taken to the preparation room. One drop of proparacaine was instilled into both eyes of the infants before the examination. Proparacaine-containing drops are used to provide topical anesthesia for rapid and short-term diagnostic or surgical procedures (Bashinsky, 2017). The third researcher then took the infants into the examination room and placed them on the examination table. A pulse oximetry probe was attached to the left foot of all infants.

Eye Examination Procedure

The third investigator placed the infant in a supine position and fixed the infant's head in a midline, slightly extended position. The eye examination was performed by an ophthalmologist (the fourth researcher). Each eye examination took approximately one to one and a half minutes. The groups were as follows:

Swaddling group (n=30) The third researcher swaddled each infant with its thin blanket. The swaddling involved bringing the infant's left hand close to the left buttock and wrapping it with the upper right end of the blanket. Similarly, she wrapped the baby's right hand with the upper left end of the blanket by bringing it closer to the right hip. She wrapped the baby's legs with the lower part of the blanket, ensuring that the baby's head could move freely.

White Noise Group (n=30) The third researcher turned on white noise (rain sound; link: https://www.youtube.com/watch?v=rZeM-HZeneo) before the start of the eye examination and played it to the infants until the end of the examination.

White Noise + Swaddling Group (n=30) The third researcher swaddled the infants in this group as described in the swaddling group and turned on the white noise (rain sound; link: https://www.youtube.com/watch?v=rZeM-HZeneo) before the examination started and played it to the infants until the examination was over.

Control Group (n=30) Babies in this group received care in accordance with the hospital routine. In the hospital routine, babies are examined with the clothes they are wearing during the examination, and no non-pharmacologic method is applied during the procedure.

All data collection was performed by a single outpatient nurse who was not part of the research team. This nurse works in the neonatal eye outpatient clinic and has a neonatal intensive care nursing certificate.

Data Collection Tools Infant Information and Monitoring Form The form was prepared by researchers (Baş et al., 2015; Francis, 2016; Sun et al., 2020; Turan et al., 2021) and consisted of 11 questions. The form included information about the infant's demographic characteristics, gestational age, birth weight, mode of delivery, gender, postnatal age, diet, Apgar score, oxygen therapy, and phototherapy. Additionally, T1, T2, and T3 pain scores, heart rates, and oxygen saturation levels were recorded.

The Premature Infant Pain Profile (PIPP) The pain score of the infants was evaluated using the PIPP. The Turkish validity and reliability of the scale, developed by Stevens et al. (2014), were performed by Taplak and Bayat (2019). The scale assesses seven items: gestational age, behavioral status, highest heart rate, lowest oxygen saturation value, forehead wrinkling, squinting, and widening of the wings of the nose. Each item is scored from 0 to 3 (from good to bad), with higher scores indicating greater pain. The total PIPP score ranges from 0 to 21, where 0-6 points indicate mild pain, 7-12 points indicate moderate pain, and 13-21 points indicate severe pain (Stevens et al., 2014).

Ethical Approval All procedures were conducted in compliance with the ethical standards of the Institutional and National Research Committee and within the guidelines of the Declaration of Helsinki. Approval was obtained from the institution and the ethics committee (date: October 26, 2020, number: E2-22-2419). The parents of the babies were informed about the purpose, method, and other details of the study. They signed a written consent form before the study commenced.

Statistical Analysis Statistical analyses were performed using the SPSS (version 27, IBM) package program. Descriptive statistics were used to interpret the findings. "Pearson-χ2" cross-tabulations were employed to examine the relationship between two qualitative variables. For normally distributed data, the "ANOVA" test (F-table value) was used to compare three or more independent groups, and the "Repeated Measures" test (F-table value) was used to compare three or more dependent groups. For non-normally distributed data, the "Kruskal-Wallis H" test (χ2-table value) was used to compare three or more independent groups, and the "Friedman" test (χ2-table value) was used to compare three or more dependent groups.

ELIGIBILITY:
Inclusion Criteria:

* infants with a gestational age of >37 6/7 weeks,
* birth weight ≥2000 g,
* 5th minute Apgar score ≥7,
* aged 30-36 days postpartum,
* undergoing their first eye examination

Exclusion Criteria:

* a history of hospitalization in the neonatal intensive care unit,
* postnatal resuscitation,
* presence or suspicion of a congenital and/or genetic disease,
* hearing problems, surgical operation for any reason,
* systemic analgesic administration within the last six hours.

Ages: 30 Days to 36 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
The Premature Infant Pain Profile total pain score | Eye examination beginning and end (approximately 1-1.5 minutes)
  The Premature Infant Pain Profile (PIPP); The scale assesses seven items: gestational age, behavioral status, highest heart rate, lowest oxygen saturation value, forehead wrinkling, squinting, and widening of the wings of the nose. Each item is scored from 0 to 3 (from good to bad), with higher scores indicating greater pain. The total PIPP score ranges from 0 to 21, where 0-6 points indicate mild pain, 7-12 points indicate moderate pain, and 13-21 points indicate severe pain
heart rate value | Eye examination beginning and end (approximately 1-1.5 minutes)
oxygen saturation value | Eye examination beginning and end (approximately 1-1.5 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Güner Başara, Dr, Study Director — Tokat Gaziosmanpaşa University Erbaa Faculty of Health Sciences, Department of Child Health and Diseases, Tokat, Türkiye; Hüsniye Çalışır, Prof. Dr., Principal Investigator — Aydın Adnan Menderes University Faculty of Nursing Child Health and Diseases Nursing , Aydın, Turkey; Emel Bahadır Arsu, Nurse, Principal Investigator — Department of Ophthalmology, Ankara Bilkent City Hospital, University of Health Sciences, Ankara, Turkey; Özdemir Özdemir, Prof. Dr., Principal Investigator — Department of Ophthalmology, Ankara Bilkent City Hospital, University of Health Sciences, Ankara, Turkey
Locations (1):
- Sultan Güner Başara, Tokat Province, Erbaa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no web address with additional information about the IPD sharing plan